CLINICAL TRIAL: NCT02539264
Title: Impact of Smoking, BZD and Obesity on Severe Obstructive Sleep Apnea (sOSA)
Brief Title: Impact of Smoking, Benzodiazepine (BZD) Use and Obesity on Severe Obstructive Sleep Apnea (sOSA)
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, FCCP, MD, FCCP, Astes
Other Study IDs: DEES-OSA
Record Dates: First submitted 2015-08-29; First posted 2015-09-03 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Obstructive Sleep Apnea; Obesity; Smoking
Keywords: All patients registered for A PSG; polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity; Smoking | interventions — Smoking Devices; Adiposity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Smoking — Influence of smoking on parameters derived from overnight PSG
Other: Obesity — Influence of obesity on parameters derived from overnight PSG
Other: Benzodiazepine use — Influence of benzodiazepine use on parameters derived from overnight PSG

SUMMARY:
In this study the investigators will analyze the influence of smoking, benzodizepine use, and obesity among patients with severe Obstructive Sleep Apnea (sOSA).

DETAILED DESCRIPTION:
This study is a retrospective study. Patients enrolled: all patients with a PSG (polysomnography) between 1st January 2014 and 30th June 2015.

First analysis: influence of smoking, benzodiazepine use, and obesity on the AHI (Apnea Hypopnea Index: the number of apnea and hypopnea per hour of sleep).

Second analysis: only among patients with sOSA: influence of smoking, benzodiazepine use, and obesity on sleep fragmentation and night oximetry.

ELIGIBILITY:
Inclusion Criteria:

* All patients registered for an overnight PSG at Clinique Saint-Luc of Bouge

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients registered for an overnight PSG at Clinique Saint-Luc of Bouge
Sampling Method: Non-Probability Sample
Enrollment: 920 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | 1 day
  Apnea Hypopnea Index (AHI) is defined as the number of apnea and hypopnea per hour of sleep. It is the major determinant of the severity of OSA.

SECONDARY OUTCOMES:
Sleep fragmentation defined by the percentage of time spent in each of the four stades of sleep (Stade 1, Stade 2, Slow wave sleep and Rapid Eye Movements) | 1 day
  Are smoking and/or obesity a risk factor for sleep fragmentation?
Time spent under 90% of SpO2 during the night | 1 day
  Are smoking and/or obesity a risk factor for oxygen desaturation (< 90% SpO2) during the night?

CONTACTS AND LOCATIONS:
Overall Officials: Eric DEFLANDRE, MD, FCCP, Principal Investigator — Astes